CLINICAL TRIAL: NCT02356250
Title: A Pilot Study: Defining Peripheral Endothelial Function in Portal Hypertensive
Brief Title: A Pilot Study: Defining Peripheral Endothelial Function in Portal Hypertensive Cirrhotic Patients
Status: Withdrawn | Type: Observational
Why Stopped: no participants enrolled
Sponsor: Eyal Ashkenazi (Other)
Responsible Party: Sponsor-Investigator, Eyal Ashkenazi, M.D, Carmel Medical Center
Organization: Carmel Medical Center (Other)
Other Study IDs: CMC 14-0117-CTIL
Record Dates: First submitted 2015-01-25; First posted 2015-02-05 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Portal Hypertension; Cirrhosis
Keywords: liver biopsy f 4
MeSH Terms: conditions — Hypertension, Portal; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PORTAL HYPERTENSION: PAIEBT WITH PORTAL HYPERTENSION

SUMMARY:
Rationale for the study:

To try and define PEF in cirrhotic patients with CSPH, and maybe to try to find a correlation between HVPG ( hepatic vein pressure gradient ) result and PEF result in a way that the result of the PEF test will be able to predict if a patient has CSPH (yes of no). By this, to try and develop a portable office-based device that can produce immediate results in a non-invasive manner in cirrhotic patients and help in evaluating prognosis in these patients in a noninvasive manner.

Aim:

The aim of this study is to try and characterize the peripheral endothelial function (PEF) in patient with cirrhosis and CSPH. This will be evaluated by measuring the PEF in every patient before evaluating his HVPG level in a hemodynamic study.

DETAILED DESCRIPTION:
To try and define PEF in cirrhotic patients with CSPH, and maybe to try to find a correlation between HVPG result and PEF result in a way that the result of the PEF test will be able to predict if a patient has CSPH (yes of no). By this, to try and develop a portable office-based device that can produce immediate results in a non-invasive manner in cirrhotic patients and help in evaluating prognosis in these patients in a noninvasive manner

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years old (Male/Female) and not more than 75 years old
2. Diagnosis of cirrhosis:

i. By liver biopsy ii. Or strong suspicion of cirrhosis by accepted criteria for the clinical diagnosis of cirrhosis (e.g. peripheral edema or varices, palpable hard left lobe of the liver, small right lobe span or palpable splenomegaly), and/or radiological evidence of cirrhosis (by abdominal US, CT, or MRI, showing a nodular liver and/or portosystemic collaterals with portal vein patency and/or ascites and/or splenomegaly, and/or colloid shift on a colloid-isotope liver-spleen scan), and/or laboratory variables (platelets <100,000/mm3, albumin< 3.5g/dL, or INR >1.3) and/or presence of esophageal varices (without previous variceal bleeding episode) or HVPG≥12mmHg from previous testing, or by FIbroscan or Fibrotest results showing fibrosis stage- 4.

c. Has been scheduled for hemodynamic study testing. d. Patients should have a Child Pugh score A or higher

Exclusion Criteria:

1. Patients already receiving beta blockers
2. Hepatocellular carcinoma
3. Portal vein thrombosis
4. Cholestatic liver disease
5. Severe heart, pulmonary or renal disease.
6. Patients with Ischemic heart disease
7. Patients with diabetes mellitus
8. Any major surgery in the past 3 months.
9. Patient is a recipient of any organ transplant
10. Patient, based on the opinion of the investigator, should not be enrolled into this study.
11. Patients unable or unwilling to sign informed consent
12. Patients that are participating in other clinical trials evaluating experimental treatments or procedures or have participated in a clinical trial in the past 3 months.
13. Active smoking
14. Uncontrolled hypertension

Withdrawal criteria:

1. Patient that based on the opinion of the investigator should be withdrawl from the study due to no compliance
2. Patient wish to stop participate in study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A maximum of 30 patients with cirrhosis Ages between 18 to 75
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-29 (Actual)

PRIMARY OUTCOMES:
is to try and characterize the peripheral endothelial function (PEF) in patient with cirrhosis and CSPH (by measuring the PEF in every patient before evaluating his HVPG level in a hemodynamic study) | 2 month for each patient and 1 year total
  by measuring the PEF in every patient before evaluating his HVPG level in a hemodynamic study

CONTACTS AND LOCATIONS:
Overall Officials: EYAL ASHKENAZI, DR, Principal Investigator — Carmel Medical Center